CLINICAL TRIAL: NCT06240949
Title: Comparative Effects of Positional Release and Manual Pressure Techniques of Tight Hip Flexors on Pain, Range of Motion, Lumbosacral Angle, and Disability in Patients With Chronic Low Back Pain
Brief Title: Comparison of Positional Release and Manual Pressure Technique in Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHs/23/0168
Record Dates: First submitted 2023-12-26; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Chronic Low-back Pain
Keywords: Low back pain; Chronic low back pain; Hip flexors; positional release technique; Manual Pressure Technique
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positional release technique (Experimental): Positional release technique will be applied on iliopsoas muscle.
  Interventions: Device: Positional Release Technique
- Manual pressure technique (Experimental): Manual pressure technique will be applied on iliopsoas muscle.
  Interventions: Device: Manual Pressure Technique

INTERVENTIONS:
Device: Positional Release Technique — Positional Release Technique will be applied on iliopsoas muscle. Treatment time will be 30 minutes per session, 4 times/week for 4 weeks in the hospital setting.
  Arms: Positional release technique
Device: Manual Pressure Technique — Manual Pressure Technique will be applied on iliopsoas muscle. Treatment time will be 30 minutes per session, 4 times/week for 4 weeks in the hospital setting.
  Arms: Manual pressure technique

SUMMARY:
The purpose of the study is to compare the effect of positional release technique and manual pressure technique of hip flexors on pain, range of motion, lumbosacral angle and disability in patients with chronic low back pain

DETAILED DESCRIPTION:
This will be Randomized clinical trial. Individuals who met inclusion criteria will be included in this study. All participants will go through randomization and divided into two groups. Pre intervention assessment is made for both groups. Then intervention will apply to both groups. Group A will receive positional release technique and Group B will be treated by manual pressure technique and pain, range of motion, lumbosacral angle and functional disability will be measured before and after the treatment using NPRS, Inclinometer and ODI. Estimated time of treatment protocol will be 30 minutes per session, 4 times/week for 4 weeks in the hospital setting. Subjects will be evaluated at baseline and 4th week assessment will be the final.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* age group 25 to 40yrs
* Atraumatic chronic low back pain more than 3 months
* Patients with Anterior pelvic tilt
* Patients with lumbosacral angle > than 50 degrees

Exclusion Criteria:

* Pregnancy
* history of vertebral fracture
* History of any spinal surgery
* Disc disease
* Osteoporosis
* Bone disease
* Patient unable to give consent

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-02-05 (Estimated); Study Completion 2024-02-05 (Estimated)

PRIMARY OUTCOMES:
Hip flexors tightness | 4th week
  Hip flexors tightness will be assessed using an inclinometer to measure the range of motion (ROM) for active hip extension and Lumbosacral angle
Pain Intensity | 4th week
  Pain intensity will be evaluated using the Numeric Pain Rating Scale (NPRS)
Functional disability | 4th week
  Functional disability will be assessed by Oswestry disability questionnaire.
Anterior pelvic tilt | 4th week
  Anterior pelvic tilt will be measured using an inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, phD, Principal Investigator — Riphah International University, Lahore; Faiza Alzaf, Principal Investigator — Riphah International University, Lahore
Locations (1):
- DHQ and tertiary hospitals, Khanewal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juker D, McGill S, Kropf P, Steffen T. Quantitative intramuscular myoelectric activity of lumbar portions of psoas and the abdominal wall during a wide variety of tasks. Med Sci Sports Exerc. 1998 Feb;30(2):301-10. doi: 10.1097/00005768-199802000-00020. PMID 9502361
- [Background] Avrahami D, Potvin JR. The clinical and biomechanical effects of fascial-muscular lengthening therapy on tight hip flexor patients with and without low back pain. J Can Chiropr Assoc. 2014 Dec;58(4):444-55. PMID 25550670
- [Background] Aslan H, Buddhadev HH, Suprak DN, San Juan JG. ACUTE EFFECTS OF TWO HIP FLEXOR STRETCHING TECHNIQUES ON KNEE JOINT POSITION SENSE AND BALANCE. Int J Sports Phys Ther. 2018 Aug;13(5):846-859. PMID 30276017
- [Background] Hoy D, Brooks P, Blyth F, Buchbinder R. The Epidemiology of low back pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):769-81. doi: 10.1016/j.berh.2010.10.002. PMID 21665125
- [Background] Naik Prashant P, Anand H, Khatri Subhash M. Comparison of muscle energy technique and positional release therapy in acute low back pain-RCT. Physiotherapy and Occupational Therapy. 2010;32
- [Background] Deyo RA, Von Korff M, Duhrkoop D. Opioids for low back pain. BMJ. 2015 Jan 5;350:g6380. doi: 10.1136/bmj.g6380. PMID 25561513
- [Background] Gonzalez-Galvez N, Gea-Garcia GM, Marcos-Pardo PJ. Effects of exercise programs on kyphosis and lordosis angle: A systematic review and meta-analysis. PLoS One. 2019 Apr 29;14(4):e0216180. doi: 10.1371/journal.pone.0216180. eCollection 2019. PMID 31034509
- [Background] Santaguida PL, McGill SM. The psoas major muscle: a three-dimensional geometric study. J Biomech. 1995 Mar;28(3):339-45. doi: 10.1016/0021-9290(94)00064-b. PMID 7730392
- [Background] Licciardone JC, Kearns CM, Crow WT. Changes in biomechanical dysfunction and low back pain reduction with osteopathic manual treatment: results from the OSTEOPATHIC Trial. Man Ther. 2014 Aug;19(4):324-30. doi: 10.1016/j.math.2014.03.004. Epub 2014 Mar 18. PMID 24704126
- [Background] Chaitow L. Positional Release Techniques E-Book: Elsevier health sciences; 2007
- [Background] Ibraheem EEMAE. Conventional therapy versus positional release technique in the treatment of chronic low back dysfunction. Int J Physiother Res. 2017;5(5):2325-31
- [Background] Hanson P, Magnusson SP, Simonsen EB. Differences in sacral angulation and lumbosacral curvature in black and white young men and women. Acta Anat (Basel). 1998;162(4):226-31. doi: 10.1159/000046437. PMID 9831771
- [Background] Mosner EA, Bryan JM, Stull MA, Shippee R. A comparison of actual and apparent lumbar lordosis in black and white adult females. Spine (Phila Pa 1976). 1989 Mar;14(3):310-4. doi: 10.1097/00007632-198903000-00011. PMID 2711246
- [Background] Naik MS, Shah DN. Prevalence of tightness in hip joint muscles in middle aged women engaging in prolonged desk job: Descriptive study. Age. 2022;43:6.077908
- [Background] AWATEF ML, ALI FAM, SHIMAA T, MAGDA GS. Effect of lumbar hyperlordosis correction on craniovertebral angle in low back pain patients. The Medical Journal of Cairo University. 2020;88(December):2051-7.